CLINICAL TRIAL: NCT05889078
Title: The Effects of Walking in Nature (vs. an Urban Setting) on the Wellbeing of Postsecondary Students.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Marie-Claude Geoffroy, Dr Marie-Claude Geoffroy, assistant professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IUSMD-18-33 Phase 2
Record Dates: First submitted 2023-05-17; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Affect; Wellness, Psychological; Depressive Symptoms; Anxiety Disorders and Symptoms; Stress; Sleep; Non-suicidal Self-injury
Keywords: Positive affect; Negative affect; Wellbeing; Walking intervention (nature vs urban); Postsecondary students; Young adults; Stress; Sleep quality; Non-suicidal self-injury; Mindfulness
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders; Self-Injurious Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature condition (Experimental): Participants will walk in a nature setting 3x per week for a period of 4 weeks.
  Interventions: Behavioral: A 4-week walking intervention
- Urban condition (Experimental): Participants will walk in an urban setting 3x per week for a period of 4 weeks.
  Interventions: Behavioral: A 4-week walking intervention

INTERVENTIONS:
Behavioral: A 4-week walking intervention — Participants will walk along a predetermined route 3 times per week for a period of 4 weeks, answering a pre- and post-intervention questionnaire as well as weekly questionnaires measuring their affect and other variables related to wellbeing. Participants will be randomly assigned to one of two conditions (nature vs urban setting), determining whether the predetermined route they will walk is in a nature or urban setting.

SUMMARY:
The goal of this randomized controlled trial is to examine the effects of a walking intervention (3 walks per week for a period of 4 weeks) in a nature vs. urban setting on the wellbeing of young adult postsecondary students. We will examine changes in positive and negative affect for participants assigned to the nature condition vs those assigned to the urban condition (primary outcome). We will also examine changes in reported depression and anxiety symptoms, perceived stress levels, sleep quality, mindfulness and wellbeing (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-25 years
* speaks English
* had working smartphone that can track walk routes using a smartphone application

Exclusion Criteria:

* inability to walk for 45 minutes due to serious medical reasons (eg surgery)
* heart condition

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline positive affect at 4 weeks | 4 weeks (1x per week for 4 weeks)
  Measured by the Positive and Negative Affect Schedule. Total scores range from 10-50 for positive affect, with higher scores indicating higher levels of positive affect (a better outcome).
Change in baseline negative affect at 4 weeks | 4 weeks (1x per week for 4 weeks)
  Measured by the Positive and Negative Affect Schedule. Total scores range from 10-50 for negative affect, with higher scores indicating higher levels of negative affect (a worse outcome).

SECONDARY OUTCOMES:
Change in baseline depression symptoms at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the Patient Health Questionnaire-9 Items (PHQ-9), with total scores ranging from 0-27, with higher scores indicating more depressive symptoms (a worse outcome).
Change in baseline anxiety symptoms at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the General Anxiety Disorder-7 (GAD-7), with total scores ranging from 0-21, with higher scores indicating greater severity in anxiety symptoms (a worse outcome).
Change in baseline perceived stress levels at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the Perceived Stress Scale (PSS), with total scores ranging from 0 to 40 with higher scores indicating higher perceived stress (a worse outcome).
Change in baseline sleep quality at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the Pittsburgh Sleep Quality Index (PSQI), with total scores ranging from 0 to 21 with higher scores indicating worse sleep quality (a worse outcome).
Change in baseline mindfulness at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the Five Facets of Mindfulness Questionnaire (FFMQ). Each item is rated from 1 = rarely true to 5 = always true. Results comprise a total average score and 5 subscale scores. Average scores are calculated by summing the responses and dividing by the number of items. Higher scores indicate higher levels of mindfulness (a better outcome).
Change in baseline levels of wellbeing at 5 weeks | 5 weeks (1 week following completion of study intervention)
  Measured by the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS), with scores ranging from 14 to 70. Higher scores indicate greater positive mental wellbeing (a better outcome).
Change in baseline non-suicidal self-injury at 5 weeks | 5 weeks (1 week following completion of study intervention)
  We assessed Non-Suicidal Self-Injury using a question previously used with same-aged participants in the Québec Longitudinal Study of Child Development: "Sometimes, some people hurt themselves intentionally, even when they don't have the intention to kill themselves. Over the past two weeks, have you harmed yourself deliberately, without the intention to kill yourself?" rated from 1 = never to 4 = very often. High scores indicate greater frequency of non-suicidal self-injury (a worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided